CLINICAL TRIAL: NCT06403904
Title: Assessing Clinical Features and Outcome of Breast Cancer in PALB2
Brief Title: Assessing Clinical Features and Outcome of Breast Cancer in PALB2 Mutation Carriers: the Palbreast Study
Acronym: PALBREAST
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, CORTESI LAURA, Principal Investigator, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: PALBREAST
Record Dates: First submitted 2023-12-22; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — An academic HRD test performed with Illumina will be performed both on PALB2-mutated and control samples. HRD will be calculated using whole-genome sequencing (WGS) data at low coverage (0.4-0.8×) for each sample using six different integrated models encompassing variable sliding windows spanning 5-1000 Kb.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male and female participants with PALB2-related BC and at least 18 years of age
- Patient affected by BC negative for mutations: The control group will be composed by patients affected by BC tested with multigene panel and resulted negative for mutations.

SUMMARY:
The Modena hereditary breast cancer group identified 3498 BRCA test candidates affected by breast cancer (BC). Among those, 392 were BRCA1/2 positive (11.2%). Since 2018, the site started to analyze eligible BC patients by multi gene panel (MGP) test. Fifty hundred sixty BRCA negative patients have been recalled, whereas other 934 were firstly analyzed by MGP. Totally, among 1494 BC patients analyzed by MGP test, 33 were PALB2 mutation carriers (2%). By involving the Italian Society of Genetic Oncology and 11 European Institutions, it is calculated to identify about 300 PALB2 mutation carriers.

PALB2 is a breast cancer susceptibility gene that encodes the BRCA2- interacting protein. Mono-allelic mutations of PALB2 are associated with an increased risk for breast and ovarian cancer in women, prostate cancer in men, and pancreatic cancer in both gender. Women with no family history of breast cancer have a cumulative risk of 33%, compared to 58% in women with two or more family members with breast cancer. Several studies with populations ranging from to 54 to 362 individuals aimed to describe breast cancer phenotypic characteristics in PALB2 mutation carriers. Some of these studies suggested an association with triple-negative phenotype, older age at diagnosis (>30 years), tumor size > 2 cm, negative HER2 status, lymph nodes positive and bilaterality. Nevertheless, results among different studies are contradictory and no data on prognosis of these patients are reported. Furthermore, the clinical potential of PARP inhibition beyond currently approved indications to additional patients whose tumors have (epi)genetic changes affecting homologous recombination repair raises new interest in PALB2 mutations as molecular target.

Primary objectives is to study the incidence and mortality rates of gPALB2 Breast Cancer.

DETAILED DESCRIPTION:
This is a multicenter hospital-based retrospective cohort control study conducted across several Institutions with known expertise in managing hereditary breast cancer.

It is planned to enrol at least 300 PALB2-related BC diagnosed at the different Units and 300 BC as control group tested for multigene panel and resulted negative for mutations. It is expected to complete the accrual in one year; furthermore, a minimum follow-up of one more year is required for the final analysis of primary and secondary endpoints.

Since some delay in the Ethical committee approvals at different Centers can rising, the study could be extended for another year Subjects will be inserted in the registry after having identified a pathogenic or likely pathogenic germline PALB2 mutation. All BC stages at the diagnosis will be included in the analysis. The BC mutation negative control group will be consecutively selected from each center, as ratio 1:1 in respect with the number of gPALB2 mutated patients enrolled, matching those for age, stage and period of diagnosis. The following data for each patient will be collected

* Demographic and clinical characteristics: age at diagnosis, BMI.
* Tumor characteristics: breast imaging (US, mammogram, breast MRI), cito-histological examination from FNA/core biopsy, multifocality or bilaterality, clinical stage at diagnosis.
* Data about surgery and pathological features: date of surgery (the date of the primary tumor removal), type of surgery, tumor size and number of positive lymph nodes (pTN), biological features on surgical sample (histological type, ER, PR, HER2, Ki-67, grade, TILs, AR).
* Systemic treatment modalities (neoadjuvant, adjuvant, advanced therapies) with a detailed description of the treatment regimens: drugs administered, dosage of drugs and duration with start and end dates. In patients that underwent neoadjuvant treatment, data about pathological response (ypTN) and local regional treatment after NAC were collected. pCR is defined as documented CR to NAC and/or ypT0/is N0.
* Type of radiotherapy performed and duration.
* Type of first relapse (local/distant), location of lesions, date of detection and therapie
* Data concerning family history and other primary tumours
* Outcomes in terms of OS and DFS.
* Patient's participation in previous studies. Patients' characteristics and the distribution of each parameter across will be reported as absolute and percentage frequencies. For each group of patients registered at different Centers, the number of all tests performed will be reported, as denominator, in order to establish the frequencies of mutations in all the European countries.

Outcomes of interest will be DFS, DDFS and OS in the cohort and control groups. DFS, DDFS and OS curves will be conducted using Kaplan-Meier method and time time-to-event distributions will be compared with log-rank test (univariate regression). Log-rank test will be used to compare the difference between values over and under the selected cut-off on survival curves. Multivariate analysis will be conducted using Cox proportional hazard models to identify significant predictors of mortality. In case of documented PD, each participant will be contacted by telephone every 12 weeks (+-14 days) to assess for survival status until withdrawal of consent to participate in the study, becoming lost to follow up, death or end of the study, whichever occurs first. Statistical analysis will be conducted using SPSS Statistics for Windows Version 23.0 (IBM Corporation, Armonk, NY, USA).

In order to minimise bias on the subjects' selection, the analysts will not be informed about the origin of the patients, being the number attributed to each centre blinded for the cohort and control group.

For details on what is included in the efficacy and safety endpoints, see Section 3 Objectives and Endpoints.

ELIGIBILITY:
Inclusion Criteria:

- 1. Has a histologically or cytologically confirmed breast cancer 2. Has any stage of BC 3. Has documented mutation in PALB2 gene (germline or somatic) that is predicted to be deleterious or suspected deleterious.

4. Has a multigene test performed and resulted negative for alterations. 5. Has information on tumours characteristics, modality of diagnosis, type of surgical treatment, medical therapy, family history and eventually second primary tumours

Demographics Is male or female, who is at least 18 years of age at the time of signing the informed consent.

Exclusion Criteria:

Has a benign variant of PALB2 gene or variant of uncertain (or unknown) significance (VUS) Is involved in the planning and/or conduct of the study Is judged by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female participants with PALB2-related BC and at least 18 years of age will be enrolled in this study. The control group will be composed by patients affected by BC tested with multigene panel and resulted negative for mutations.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this trial is to evaluate the frequency of PALB2-related BC in the different European countries, reflecting the real needs for this patients' population. | 36 months
  The main objective is to evaluate the frequency of PALB2-related BC in the different European countries, reflecting the real needs for this patients' population.

CONTACTS AND LOCATIONS:
Overall Officials: LAURA CORTESI, MD, Principal Investigator — Azienda Ospedaliero Universitaria Policlinico Modena
Locations (1):
- Aou Modena, Modena, Italy